CLINICAL TRIAL: NCT07000786
Title: EUmetriosis: Insights Into the Pathogenesis of Endometriosis
Acronym: EUmetriosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EUmetriosis
Record Dates: First submitted 2025-05-12; First posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-06

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis | interventions — Menstrual Hygiene Products; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Epigenetics characterization (Experimental)
  Interventions: Procedure: Endometrial biopsy or menstrual cup and blood sample

INTERVENTIONS:
Procedure: Endometrial biopsy or menstrual cup and blood sample — Enrolled patients will give their menstrual effluent either via a menstrual cup or via a pipelle biopsy. They will also undergo a blood draw.

SUMMARY:
This study investigates epigenetic changes in menstrual effluent and plasma from women with endometriosis to identify potential non-invasive diagnostic biomarkers for the disease.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal
* In spontaneous menstrual cycle (no hormonal treatments for the last 3 months)
* Healthy or with a clear diagnosis of endometriosis via ultrasound, MRI or laparoscopy

Exclusion Criteria:

* HIV or Hepatitis positive
* Pregnancy

Ages: 18 Years to 56 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Epigenetic analysis | Throughout the entire study, approximately during 3,5 years
  Histone post-translational modifications
Epigenetic analysis | Throughout the entire study, approximately during 3,5 years
  miRNA

CONTACTS AND LOCATIONS:
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No